CLINICAL TRIAL: NCT01130779
Title: The Continuation of Erlotinib Treatment in Non-small Cell Lung Cancer Patients Whose Brain Lesion is the Only Site of Progression : Pilot Study
Brief Title: The Continuation of Erlotinib
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Samsung Medical Center (Other)
Responsible Party: Myungju Ahn Ph.D., M.D., Samsung Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2009-07-078
Record Dates: First submitted 2010-05-25; First posted 2010-05-26 (Estimated); Last update posted 2010-05-26 (Estimated); Status verified 2010-05

CONDITIONS: Non-small Cell Lung Cancer
Keywords: Non-small Cell Lung Cancer; Erlotinib; brain metastasis
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Brain Neoplasms | interventions — Erlotinib Hydrochloride

ARMS (1):
- tarceva (Experimental): continuation of tarceva
  Interventions: Drug: Erlotinib (TARCEVA®)

INTERVENTIONS:
Drug: Erlotinib (TARCEVA®) — Erlotinib 150mg/day, everyday

SUMMARY:
Newly developed or progressive brain metastasis during erlotinib treatment is considered progressive disease requiring change of treatment regimens despite no progression in extracranial lesions. Given that there is a dissociation in terms of response to erlotinib between brain and extracranial sites, we intend to conduct this pilot study to determine whether the continuation of erlotinib treatment can prolong the progression free interval of extracranial lesions as long as cranial lesion is controlled separately by conventional treatment modalities such as surgical resection, stereotactic radiosurgery, and whole brain radiotherapy.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically or cytologically proven non small cell lung cancer
2. New developed or progression of brain lesions among patients with good control of extracranial lesions to erlotinib
3. patients who are receiving erlotinib as salvage therapy
4. At least one unidimensionally measurable lesion with a diameter > 10mm using brain MRI
5. at least on unidimensionally measurable or evaluable lesion
6. male or female patients aged >18 years
7. ECOG performance status 0-2
8. Adequate hematologic function
9. adequate renal function
10. adequate hepatic function

Exclusion criteria

1. leptomeningeal metastases
2. acute severe infection requiring antibiotic therapy
3. significant cardiovascular disease
4. uncontrolled DM
5. severe ophthalmologic disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Estimated)
Dates: Start 2009-08; Primary Completion 2010-08 (Estimated)

PRIMARY OUTCOMES:
progression free survival | 6 months

SECONDARY OUTCOMES:
overall survival | 6 months
response rate | 6 months
time to treatment failure | 6 months
toxicity profiles | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Myungju Ahn, Ph.D., M.D., Principal Investigator — Samsung Medical Center
Locations (1):
- Samsung Medical Center, Seoul, South Korea